CLINICAL TRIAL: NCT00732875
Title: A Placebo-controlled, Double-blinded, Randomized Clinical Trial of Anti-TNF Chimeric Monoclonal Antibody (cA2) in Korean Patients With Active Rheumatoid Arthritis Despite Methotrexate Treatment (Open-label Extension Part)
Brief Title: A Trial of Anti-TNF Chimeric Monoclonal Antibody (cA2) in Korean Patients With Active Rheumatoid Arthritis Despite Methorexate (Extension Part)(Study P05645)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05645
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Infliximab + Methotrexate (Experimental): Open label Infliximab infusions at weeks 0, 2, and 6 and every 8 weeks + methotrexate (MTX)
  Interventions: Biological: Infliximab + methotrexate (MTX)

INTERVENTIONS:
Biological: Infliximab + methotrexate (MTX) — Open label Infliximab infusions at weeks 0, 2, and 6 and every 8 weeks + methotrexate (MTX)
  Other Names: Remicade; SCH 215596

SUMMARY:
This trial is extension part of the P04280 (placebo-controlled, double-blind, randomized study of chronic treatment with infliximab in approximately 140 patients, NCT00202852). This study will be conducted at 6 study centers in South Korea. After completion of the last follow-up visit at Week 30 and code break in main double-blind trial, subjects randomized to the placebo group and those who were treated with an infliximab-containing regimen who maintained clinical response at the time of study completion will be provided with open-label infliximab for treatment of their conditions and additional safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients received placebo in main double-blind study (P04280, NCT00202852)
* Patients received Infliximab-containing regimen showing clinical response at week 30 in main double-blind study (P04280)

[Main double-blind study (P04280, NCT00202852) inclusion criteria]

* Diagnosis of rheumatoid arthritis (RA) according to the revised 1987 criteria of the American Rheumatism Association (Arnett et al, 1988). The disease should have been diagnosed >6 months prior to screening.
* Active disease at the time of screening and pre-infusion as defined by:

  * >=6 swollen joints
  * >=6 tender joints and
* 2 of the following:

  * morning stiffness >=45 min
  * erythrocyte sedimentation rate (ESR) >=28 mm/h
  * C-reactive protein (CRP) >=20 mg/L
* Men and women, >=18 to <=75 years of age
* Men and women of childbearing potential must be using adequate birth control measures (abstinence, oral contraceptives, intrauterine device (IUD), barrier method with spermicide, or surgical sterilization) and should continue such precautions for 6 months after receiving the last infusion.
* Must have been using oral or parenteral MTX for >3 months with no break(s) in treatment of >2 weeks total during this period. Patients must have been on a stable dose of >=12.5 mg/wk (maximum 20 mg/wk) for at >4 weeks prior to screening.
* Must be on a stable dose of folic acid prophylaxis for >4 weeks prior to screening.
* Patients using oral corticosteroids, must have been on a stable dose of <=10 mg/day for >4 weeks prior to screening. If currently not using corticosteroids the patient must have not received corticosteroids for >4 weeks prior to screening.
* If using nonsteroidal anti-inflammatory drugs (NSAIDs), patients should have been on a stable dose for >4 weeks prior to screening.
* The screening laboratory tests must meet the following criteria:

  * Hemoglobin >=5.3 mmol/L (>=8.5 g/dL), providing a low hemoglobin level is not due to nutritional deficiencies or due to diseases other than chronic RA
  * white blood cell (WBC) >=3.5 x 10^9/L (>=3.5 x 10^3/mm^3)
  * Neutrophils >=1.5 x 10^9/L (>=1.5 x 103/mm^3)
  * Platelets >=100 x 10^9/L (>=100 x 103/mm^3)
  * Serum transaminase <=2 times the upper limit of normal
  * Alkaline phosphatase levels <=2 times the upper limit of normal
  * Serum creatinine <=150 µmol/L (<=1.7 mg/dL)
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Must be capable of giving informed consent and the consent must have been obtained prior to any study procedures including wash-out period.

Exclusion Criteria:

* Exclusion criteria below of main double-blind study (P04280, NCT00202852)

[Main double-blind study (P04280, NCT00202852) exclusion criteria]

* Pregnant women, nursing mothers, or a planned pregnancy within 1.5 years of enrollment.
* Patients who are incapacitated, largely or wholly bedridden or confined to a wheelchair, and who have little or no ability for self-care.
* Patients who have any current systemic inflammatory condition with signs and symptoms that might confound the evaluations of benefit from infliximab, eg Lyme disease, or a rheumatic disease other than RA.
* Use of disease modifying anti-rheumatic drugs (DMARDs) other than MTX within 4 weeks prior to screening. (If a patient had prior exposure to leflunomide within the past 6 months, cholestyramine 8 g should be given 3 times daily for 11 days to rapidly lower the plasma level of leflunomide.)
* Use of intra-articular, i.m. or i.v. corticosteroids (including i.m. ACTH) within 4 weeks prior to screening.
* Have been previously treated with infliximab or genetic recombinant therapy with RA (e.g. etanercept, adalimumab)
* Treatment with any other therapeutic agent targeted at reducing TNF (eg, pentoxifylline or thalidomide) within the previous 3 months.
* Treatment with any investigational drug within the previous 3 months.
* Prior use of cyclophosphamide, nitrogen mustard, chlorambucil, or other alkylating agents.
* History of any clinically significant adverse reaction to murine or chimeric proteins, including but not limited to allergic reactions.
* History of infected joint prosthesis within previous 5 years.
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months.
* Chronic infectious disease such as chronic renal infection, chronic chest infection with bronchiectasis or sinusitis.
* Active tuberculosis (TB). Also excluded are patients who have evidence of latent TB (positive purified protein derivative [PPD] skin test or a history of latent TB) without adequate therapy for TB initiated prior to first infusion of study drug. Also excluded are patients with evidence of an old or latent TB infection without documented adequate therapy, if they will not be treated with antitubercular therapy during the trial. Patients with a current close contact with an individual with active TB will also be excluded. Additionally, patients who have completed treatment for active TB within the previous 2 years are now explicitly excluded from the trial. Patients with a household member who has a history of active pulmonary TB should have had a thorough evaluation for TB prior to study enrollment as recommended by a local infectious disease specialist or published local guidelines of TB control agencies. Also excluded are patients with opportunistic infections, including but not limited to evidence of active cytomegalovirus, active Pneumocystis carinii, aspergillosis, or atypical mycobacterial infection, etc, within the previous 6 months.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
* History of lymphoproliferative disease including lymphoma or signs suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic areas), or splenomegaly.
* Any current known malignancy or history of malignancy within the previous 5 years, except for squamous or basal cell carcinoma of the skin that have been treated with no evidence of recurrence.
* Patients with moderate or severe heart failure (New York Heart Association [NYHA] class III/IV).
* Patients with pre-existing or recent onset of central nervous system demyelinating disorders.
* Known recent substance abuse (drug or alcohol).
* Patients in whom multiple venipunctures are not feasible due to poor tolerability or lack of easy access.
* Have a known infection with HIV or known active hepatitis B/C infection (including associated chronic active hepatitis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Kim J, Ryu H, Yoo DH, Park SH, Song GG, Park W, Cho CS, Song YW. A clinical trial and extension study of infliximab in Korean patients with active rheumatoid arthritis despite methotrexate treatment. J Korean Med Sci. 2013 Dec;28(12):1716-22. doi: 10.3346/jkms.2013.28.12.1716. Epub 2013 Nov 26. PMID 24339699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects showing clinical response at Week 30 of a previous double-blind study of infliximab vs placebo (P04280,NCT00202852) were eligible for this study. A total of 105 subjects were eligible (67 from previous placebo & 38 from previous infliximab group) for this extension study, among whom a total of 92 enrolled to participate in the extension.
Pre-assignment Details: Of the 92 enrolled subjects, 61 were from the placebo group and 31 from the infliximab group of the previous study.
Period: Overall Study
Arm/Group | Open Label Infliximab + Methotrexate
Started | 92
Completed | 57 (These participants continued treatment until trial was completed by Sponsor.)
Not Completed | 35
Not completed — Adverse Event | 16
Not completed — Withdrawal by Subject | 6
Not completed — Lack of Efficacy | 13

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Infliximab + Methotrexate
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.1)
Age, Customized [Number; unit: participants]
  <30 years | 2
  Between 30 and less than 40 years | 14
  Between 40 and less than 50 years | 29
  Between 50 and less than 60 years | 29
  Between 60 and less than 70 years | 15
  >=70 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Any Adverse Event
Time Frame: throughout entire study (61 +/- 28.9 weeks on average)
Population: All participants were included regardless of how long they stayed in the study.
Measure: Number; unit: participants
Arm/Group | Open Label Infliximab + Methotrexate
Number analyzed (Participants) | 92
participants | 76

2. Primary Outcome: Number of Subjects Experiencing Serious Adverse Event
Description: Serious adverse events are defined as death, life-threatening events, persistent or significant disability/incapacity, hospitalization or prolongation of hospitalization and congenital anomalies.
Time Frame: throughout entire study (61 +/- 28.9 weeks on average)
Population: All participants were included regardless of how long they stayed in the study.
Measure: Number; unit: participants
Arm/Group | Open Label Infliximab + Methotrexate
Number analyzed (Participants) | 92
participants | 12

3. Primary Outcome: Number of Subjects Experiencing Any Infection
Time Frame: throughout entire study (61 +/- 28.9 weeks on average)
Population: All participants were included regardless of how long they stayed in the study
Measure: Number; unit: participants
Arm/Group | Open Label Infliximab + Methotrexate
Number analyzed (Participants) | 92
participants | 41

ADVERSE EVENTS:
Description: During conduct of the trial, adverse events were summarized using WHOART dictionary terms. Adverse events were recoded to MedDRA terms for this section of the results display.
Arm/Group | Open Label Infliximab + Methotrexate
Serious Adverse Events (participants affected / at risk) | 12/92
Other Adverse Events (participants affected / at risk) | 50/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Infliximab + Methotrexate (N=92)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
gastric ulcer (Gastrointestinal disorders) | 1 (2)
chest discomfort (General disorders) | 1 (1)
inflammation (General disorders) | 1 (1)
infusion related reaction (General disorders) | 1 (1)
ulcer (General disorders) | 1 (1)
cholecystitis acute (Hepatobiliary disorders) | 1 (1)
anaphylactoid reaction (Immune system disorders) | 1 (1)
chronic sinusitis (Infections and infestations) | 2 (2)
pneumonia cryptococcal (Infections and infestations) | 1 (1)
pyelonephritis acute (Infections and infestations) | 1 (1)
thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
confusional state (Psychiatric disorders) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
flushing (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Infliximab + Methotrexate (N=92)
diarrhoea (Gastrointestinal disorders) | 5 (6)
nausea (Gastrointestinal disorders) | 8 (11)
vomiting (Gastrointestinal disorders) | 5 (5)
chills (General disorders) | 6 (8)
nasopharyngitis (Infections and infestations) | 6 (6)
upper respiratory tract infection (Infections and infestations) | 19 (27)
alanine aminotransferase increased (Investigations) | 6 (7)
aspartate aminotransferase increased (Investigations) | 5 (6)
headache (Nervous system disorders) | 8 (9)
cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
pruritus (Skin and subcutaneous tissue disorders) | 11 (13)
urticaria (Skin and subcutaneous tissue disorders) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed publications/presentations by the investigators or their personnel/associates resulting from/relating to this study must be submitted to SP Korea for review and approval before submission for publication/presentation. If the proposed publication/presentation contains patentable subject matter, which, at SP Korea's sole discretion, warrants intellectual property protection, SP Korea may delay any publication or presentation for the purpose of pursuing such protection.